CLINICAL TRIAL: NCT04573569
Title: Neural Correlates of Cognition and Mood
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: NEUROSURG-2019-28063
Record Dates: First submitted 2018-12-16; First posted 2020-10-05 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Epilepsy, Complex Partial
MeSH Terms: conditions — Epilepsy, Complex Partial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Behavioral testing — Patients recruited for this study have already undergone surgical implantation of invasive electrodes for purpose of localizing and characterizing electrographic seizures as part of the second phase of surgical epilepsy evaluation. Patients who consent and complete enrollment will then be asked to complete cognitive and behavioral tasks on a portable computer or tablet PC while the invasive electrodes remain implanted. Tasks typically require the patient to think or act and then respond by interacting minimally with the portable computer. These tasks are performed at the will of each patient during their stay in the intensive care unit while surgical electrodes remain.

SUMMARY:
The overall objective of this study is to determine the neural correlates of cognition and mood. This study represents the first preliminary study to begin investigating cognitive and emotional states in patients who have undergone implantation of invasive electrodes for the purpose of seizure localization. In the post-implantation paradigm where patients remain under close supervision with intracranial instrumentation for recording, this study aims to create the platform and preliminary data to inform a larger study for calibrated examination of neural correlates of cognition and mood. As such, this study has the following specific aims:

Aim 1: Establish a portable platform for the assessment of cognitive, behavioral, and emotional tasks with time synchronization to ECoG/SEEG recording platform Aim 2: Quantify the variance in clinical assessments of mood and cognitive function in patients undergoing phase II epilepsy monitoring Aim 3: Assess the relationship between validated surveys/tasks and electrophysiology

DETAILED DESCRIPTION:
Study interventions are limited entirely to validated surveys completed on a computer or tablet PC, as outlined above. Patients may elect to have electrodes to be implanted that are not used in standard-of-care at this institution, but are FDA-approved for the same indications. Patients who consent and complete enrollment will be asked to complete cognitive and behavioral tasks on a portable computer or tablet PC while the invasive electrodes remain implanted. Tasks typically require the patient to think or act and then respond by interacting minimally with the portable computer.

The primary outcome for this study includes percentage of completed cognitive or behavioral tasks as a measure of the feasibility of the administration of these tasks. As this is a feasibility study, we are interested in the practical aspects of data acquisition.

Secondary outcomes include the cognitive and behavioral tasks themselves and their relationship with electrophysiology.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to consent for themselves and the patient has or is scheduled for surgically implanted electrodes for the purposes of phase II epilepsy surgical evaluation.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing Phase II surgical epilepsy localization
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage of completed cognitive tasks | Up to 1 month (Assessments start after Post-operative day 2)
  The primary outcome for this study includes percentage of completed cognitive or behavioral tasks as a measure of the feasibility of the administration of these tasks. We are interested in the practical aspects of data acquisition. No comparison is made as no baseline data exists ECoG, SEEG recordings, and eye-tracking data are timestamped, this allows the validated surveys and tasks to be linked precisely. These results will establish the response rate to the intervention allowing calculation of the number of events to use in establishing relationships with the underlying physiology.

SECONDARY OUTCOMES:
Secondary outcomes include the cognitive and behavioral tasks themselves and their relationship with electrophysiology of the brain. | Up to 1 month (Assessments start after Post-operative day 2)
  Event-related potential will be calculated using time synchronized ECoG or SEEG recordings. Averaging will be performed across each task for event-related potentials and compared with shuffled data for bootstrapping about the median. Alpha is selected to be 0.05 with the Bonferroni correction with the number of tests. Causal inference will be used to assess the relationship between the various electrodes. Causal metrics including multivariate Granger causality and Transfer Entropy will be used to assess the adjacency matrices. Statistics are performed with shuffled bootstrapping also using the Bonferroni adjustment on the number of channels. The relationship between pupil size, gaze location, task behavior and E-phys measures will be assessed with generalized linear models, generalized canonical correlation analysis, and structured equation models.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided